CLINICAL TRIAL: NCT05878795
Title: Written Exposure Therapy for Suicide Prevention (WET-SP)
Brief Title: Written Exposure Therapy for Suicide Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-43849; W81XWH-22-1-1059 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Suicide, Attempted; Suicide Threat
Keywords: Self-injurious thoughts and behaviors (SITBs); Written Exposure Therapy for Suicide Prevention (WET-SP); Military service members; Treatment as usual (TAU)
MeSH Terms: conditions — Suicide, Attempted; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written Exposure Therapy-for Suicide Prevention (WET-SP) +TAU (Experimental): Participants randomized into this arm will be offered WET-SP which will consist of 5 treatment sessions, conducted daily while the participant is hospitalized, allowing for the largest dose of treatment possible while inpatient. If a patient is discharged prior to the completion of WET-SP, the remaining sessions will be conducted in outpatient sessions. Participants in this arm will also be offered TAU.
  Interventions: Behavioral: WET-SP; Behavioral: TAU
- Treatment as usual (TAU) (Active Comparator): Participants randomized into this arm will be offered TAU which consists of daily contact and patient centered care by the acute psychiatric inpatient unit provider team (e.g., psychiatrists, therapists, case managers, behavioral health techs). Participants will engage with the provider team daily throughout the duration of hospitalization.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: WET-SP — WET-SP will consist of 5 treatment sessions; the first session lasting about one hour and each subsequent session lasting approximately 40 minutes. Each session will include a 30-minute written exposure exercise. The participant will be given general instructions for completing the narrative writings and specific instructions for completing the first session. Participants will be instructed to write about the same suicidal crisis during each session. The therapist will emphasize the importance of delving into their deepest emotions surrounding the suicidal crisis as well as the importance of writing detailed information about the crisis. Following writing, the therapist and the participant will process the writing experience. Subsequent sessions involve the therapist iteratively providing feedback to the patient regarding their writing from the previous session.
  Arms: Written Exposure Therapy-for Suicide Prevention (WET-SP) +TAU
Behavioral: TAU — TAU includes initial psychiatric stabilization, nurse case management, medication management, psychoeducation groups, and discharge planning. Patients engage with the provider team daily throughout the duration of hospitalization and have structured times for psychoeducation groups, case management, medication management, hygiene, and meals.

SUMMARY:
Military service members admitted to inpatient psychiatry for self-injurious thoughts and behaviors (SITBs) represent an at-risk group for continued SITBs and rehospitalizations in the post-discharge period. However, there is an absence of evidence-based interventions designed to be delivered on inpatient psychiatric units to reduce the risk of post-discharge SITBs. To address this gap, the investigator's research group developed Written Exposure Therapy for Suicide Prevention (WET-SP), a brief, scalable, suicide-specific psychotherapy based on the written disclosure paradigm. Written disclosure, in which an individual writes about a personally stressful experience and the related thoughts and feelings, yields improvements across physical and psychiatric domains. Pilot data suggest that written exposure also yields reductions in SITBs. Yet, no study has adapted the written exposure paradigm specifically to target the amelioration of distress associated with suicidal crises and examined whether implementing WET-SP reduces the risk of subsequent SITBs and suicide-related hospitalizations.

The primary objective of this randomized controlled trial (RCT) is to evaluate the efficacy of WET-SP, in reducing the incidence and severity of SITBs in active duty military service members following a psychiatric hospitalization due to suicidal ideation, suicide plans, or a suicide attempt. Secondary objectives are to evaluate a potential mechanism of change (i.e., decreases in thwarted belongingness [cf. social disconnectedness]) and moderator of outcomes (i.e., arc of narrative [cf. linguistical parameters of the written narratives generated during treatment]). Participants randomized to WET-SP + TAU will receive five sessions of WET-SP delivered by the study team during their psychiatric hospitalization plus treatment-as-usual (TAU). Participants randomized to TAU will receive daily contact and patient-centered care delivered by the acute psychiatric inpatient unit provider team (e.g., psychiatrists, therapists, case managers). TAU includes psychiatric assessment, initial stabilization, nurse case management, medication management, treatment of medical comorbidities, group and individual therapy, and discharge planning. Outcome assessments will be administered at pretreatment, posttreatment, and 10-, 20-, and 30-week follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Current active duty military service member, veteran, and beneficiaries
* Admitted to Carl R. Darnall Army Medical Center (CRDAMC) for suicidal thoughts, a suicide plan, or a suicide attempt
* Elevated levels of suicidal ideation severity in the past two weeks, as indicated by a score >= 3 on the Depressive Symptom Index-Suicidality Subscale (DSI-SS)
* Ability to read, write, and speak English

Exclusion Criteria:

* Active psychosis as the priority of care for hospitalization
* Moderate or greater cognitive impairment (as determined by the inability to comprehend the baseline screening questionnaires)
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Suicidal ideation (SI) | Baseline, 10 weeks
  Measured by the Depressive Symptom Index-Suicidality Subscale (DSI-SS) which is a four-item self-report focusing on frequency and intensity of suicidal thoughts and urges during the past 2 weeks. Each item is scored on a 4-point Likert scale ranging from 0 to 3. Total scores can range from 0 to 12, with higher scores representing increased severity of suicidal ideation.
SI at 20 weeks | 20 weeks
  Measured by the Depressive Symptom Index-Suicidality Subscale (DSI-SS) which is a four-item self-report focusing on frequency and intensity of suicidal thoughts and urges during the past 2 weeks. Each item is scored on a 4-point Likert scale ranging from 0 to 3. Total scores can range from 0 to 12, with higher scores representing increased severity of suicidal ideation.
SI at 30 weeks | 30 weeks
  Measured by the Depressive Symptom Index-Suicidality Subscale (DSI-SS) which is a four-item self-report focusing on frequency and intensity of suicidal thoughts and urges during the past 2 weeks. Each item is scored on a 4-point Likert scale ranging from 0 to 3. Total scores can range from 0 to 12, with higher scores representing increased severity of suicidal ideation.

SECONDARY OUTCOMES:
Most severe SI | Baseline,10 weeks, 20 weeks, 30 weeks
  The most severe SI since the last assessment will be measured using the Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R) which is a clinical interview of the presence, frequency, and characteristics of suicide and self-harming thoughts and behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Marx, PhD, Principal Investigator — Dept of Psychiatry, Chobanian & Avedisian BU School of Medicine and VA Boston Healthcare System
Locations (1):
- University of Texas Health Center San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No